CLINICAL TRIAL: NCT03060083
Title: A Randomized Trial to Compare Switching to Very Low Nicotine Content Cigarettes vs Reducing Cigarettes Per Day
Brief Title: Switching to Very Low Nicotine Content Cigarettes vs Reducing Cigarettes Per Day
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Elias Klemperer, Predoctoral Trainee, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHRMS 16-395; P00044 (Other: Center for Tobacco Products)
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Products; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Switch to VLNC cigarettes (Experimental): Participants will be instructed to use nicotine patches and gradually switch to very low nicotine content (VLNC) cigarettes throughout the study period. They will receive regular nicotine cigarettes (16.5 mg/g) during week 1, 11.26 mg/g cigarettes during week 2, 5.54 mg/g cigarettes during week 3, 2.54 mg/g cigarettes during week 4, and 0.44 mg/g cigarettes during week 5.
  Interventions: Other: Very low nicotine content (VLNC) cigarettes and nicotine replacement therapy (NRT)
- Reduce CPD (Experimental): Participants will be instructed to use nicotine patches and gradually reduce the number of regular nicotine content cigarettes that they smoke throughout the study period. They will receive regular nicotine content cigarettes (16.5 mg/g) throughout the study study period. After establishing a baseline CPD during week 1, participants will receive 70% of their baseline CPD during week 2, 35% during week 3, 15% during week 4, and 3% during week 5. Participants will receive a minimum of 1 CPD during week 5.
  Interventions: Other: Reduce cigarettes per day (CPD) with nicotine replacement therapy (NRT)

INTERVENTIONS:
Other: Very low nicotine content (VLNC) cigarettes and nicotine replacement therapy (NRT) — Participants will switch to very low nicotine content (VLNC) cigarettes with the aid of nicotine replacement therapy (NRT)
  Arms: Switch to VLNC cigarettes
Other: Reduce cigarettes per day (CPD) with nicotine replacement therapy (NRT) — Participants will reduce cigarettes per day (CPD) with the aid of nicotine replacement therapy (NRT)
  Arms: Reduce CPD

SUMMARY:
The FDA recently gained the authority to regulate the nicotine content of cigarettes. Prior research suggests that smokers who switch to very low nicotine content (VLNC) cigarettes experience reduced addiction to nicotine and are more likely to quit smoking. Currently, the most common method for smokers to reduce their nicotine intake is to reduce their number of cigarettes per day (CPD). No research has compared reducing smokers' nicotine intake by switching to VLNC cigarettes vs by reducing CPD with regard to decreasing dependence or quitting; thus the investigators will examine the two strategies by randomizing smokers to 1) switch to VLNC cigarettes or 2) reduce CPD. In addition, all smokers will use the nicotine patch to help them reduce their nicotine intake.

DETAILED DESCRIPTION:
Primary:

1. Determine the relative feasibility of switching to VLNC cigarettes vs reducing CPD when all participants are aided by nicotine replacement therapy (NRT).
2. Determine whether switching to VLNC cigarettes or reducing CPD more effectively reduces nicotine dependence when all participants are aided by NRT.

   Secondary:
3. Determine whether switching to VLNC cigarettes vs reducing CPD increases quit attempts and 7-day point-prevalence abstinence more when all participants are aided by NRT.
4. Determine the relative effectiveness of switching to VLNC cigarettes and reducing CPD when all participants are aided by NRT with comparisons of a) craving, b) withdrawal, c) perceived harm from smoking and d) participants' enjoyment from smoking.
5. Determine whether switching to VLNC cigarettes or reducing CPD increases use of e-cigarettes or other non-combustible nicotine products more.

Rationale for Proposed Study:

A policy to reduce the nicotine content of cigarettes could be useful for the majority of smokers who are not ready to quit. Specifically, the FDA recently gained the authority to regulate cigarettes' nicotine content and switching to very low nicotine content (VLNC) cigarettes has been proposed as a future regulatory policy to give smokers the option to decrease nicotine intake from cigarettes in order to decrease nicotine dependence and quit smoking. A review of clinical trials suggest that switching to VLNC cigarettes with and without nicotine replacement therapy (NRT) reduces dependence, carcinogens, and carbon monoxide and increases quitting; however, its long-term effects are unclear.

Nicotine dependence is determined by nicotine intake (i.e., yield) as well as non-nicotine reinforcers conditioned by the repetitive act of smoking (i.e., multiple cigarettes per day). Presently, reducing cigarettes per day (CPD) is the most common strategy to reduce nicotine intake and appears to be an effective method of reducing dependence. However, a regulatory policy that introduces VLNC cigarettes will provide smokers with the opportunity to reduce nicotine intake without changing the frequency of their smoking behavior (i.e., CPD). Thus, reducing nicotine by switching to VLNC cigarettes may affect conditioned reinforcers and dependence differently than reducing nicotine intake via reducing CPD. The investigators know of no research that has compared the regulatory policy of reducing nicotine intake via VLNC cigarettes vs the common method of reducing nicotine intake via reducing CPD. This comparison will provide important information regarding the components involved in changing nicotine dependence and the potential effects of a policy that regulates the nicotine content of cigarettes.

NRT appears to increase the feasibility and effectiveness of switching to VLNC cigarettes as well as reducing full nicotine CPD. In both scenarios, NRT facilitates a net reduction in nicotine. Further, NRT is currently available to smokers who reduce CPD, will be available to smokers if cigarettes' nicotine levels are reduced by the FDA, and is likely to be used as an aid for both.

The present study will compare participants who switch to VLNC cigarettes vs participants who reduce CPD when all participants receive NRT patch. Specifically this comparison will examine differences in feasibility and effectiveness of reducing nicotine dependence.

Study Design:

Consenting participants will be randomly assigned to 1) switch to VLNC cigarettes with NRT or 2) reduce full nicotine CPD with NRT during the 5-week study period. All participants will complete baseline measures and receive full nicotine or VLNC study cigarettes as well as weekly supplies of 21-mg nicotine patches with instructions to replace their old patch with a new patch each morning.

During their first study visit, the investigators will provide all participants with a one-week supply of full nicotine study cigarettes (16.5 ± 0.17 mg/g) that totals 150% of their normal number of CPD in order to establish a baseline CPD with novel study cigarettes that are being provided free of charge. The 16.5 mg/g nicotine content NIDA research cigarette is estimated to have a nicotine yield (0.8 mg) similar to many commercial cigarettes. Participants will be instructed to smoke only study cigarettes, but to smoke as usual during the first week of the study. All study cigarettes are for investigational purposes only and are not available or intended for commercial use.

Switching to VLNC cigarettes Participants who are randomized to switch to VLNC cigarettes will receive a supply of 100% of their baseline number of CPD during study visits (determined during week 1) throughout weeks 2 to 5 and instructed to smoke as usual (e.g., not to attempt to reduce CPD). They will receive study cigarettes with progressively lower nicotine content (mg/g tobacco) beginning with 11.26 ± 0.11 mg/g during week 2, 5.54 ± 0.27 mg/g during week 3, 2.54 ± 0.05 mg/g during week 4, and 0.44 ± 0.01 mg/g during week 5. Participants will also receive a supply of NRT patches with instructions to wear one patch per day every day throughout weeks 2 through 5. This schedule was selected based on available VLNC cigarettes and findings that indicate that a gradual transition to cigarettes with a nicotine content of approximately 1 mg/g or less with the NRT patch is safe, effective and feasible. The investigators will estimate NRT use and compliance with VLNC study cigarettes with daily and weekly self report.

Reducing CPD The investigators will provide participants who are randomized to reduce CPD with full nicotine study cigarettes (16.5 ± 0.17 mg/g) during each study visit throughout the 5-week study period and instruct them to only smoke cigarettes provided by the study. After establishing a baseline CPD during week 1, participants will receive progressively fewer cigarettes beginning with 70% of their baseline CPD during week 2, 35% during week 3, 15% during week 4, and 3% during week 5. Participants will receive a minimum of 1 CPD during week 5. Participants will also receive a supply of NRT patches with instructions to wear one patch per day every day throughout weeks 2 through 5. This schedule was selected to match the percent reduction in nicotine content of cigarettes for smokers randomized to switch to VLNC cigarettes. Further, this schedule of NRT aided reductions in CPD appears to be safe, feasible and effective. The investigators will estimate reductions in CPD, compliance with study cigarettes, and NRT use with daily and weekly self-report.

ELIGIBILITY:
Eligibility will be determined based on:

* participants' age,
* their cigarettes smoked per day,
* their intention to quit,
* their willingness to use medications,
* prior use of tobacco and non-tobacco nicotine products,
* prior use of stop-smoking services or medications,
* DSM 5 criteria for Tobacco Use Disorder,
* current use of opioid maintenance medications,
* access to a telephone and the Internet,
* proximity to the University of Vermont,
* their bed time,
* status as a US citizen,
* comfort speaking, reading and writing in English, and
* whether or not the participant is breast feeding, pregnant or has the potential to become pregnant or begin breastfeeding during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klemperer EM, Hughes JR, Callas PW, Benner JA, Morley NE. Effectiveness of switching to very low nicotine content cigarettes plus nicotine patch versus reducing daily cigarette consumption plus nicotine patch to decrease dependence: an exploratory randomized trial. Addiction. 2019 Sep;114(9):1639-1650. doi: 10.1111/add.14666. Epub 2019 Jun 30. PMID 31106492
- [Result] Klemperer EM, Hughes JR, Callas PW. Increasing Quit Attempts by Transitioning to Very Low Nicotine Content Cigarettes Versus Reducing Number of Cigarettes Per Day: A Secondary Analysis of an Exploratory Randomized Trial. Nicotine Tob Res. 2019 Dec 23;21(Suppl 1):S81-S87. doi: 10.1093/ntr/ntz145. PMID 31867643
- [Result] Nighbor TD, Klemperer EM, Hughes JR, Reed EN, Simone SJ, West JC. Both reducing cigarettes per day and transitioning to very low-nicotine-content cigarettes decreases demand for usual-brand cigarettes. Exp Clin Psychopharmacol. 2021 Dec;29(6):587-592. doi: 10.1037/pha0000403. Epub 2020 Jul 13. PMID 32658536
- See also: This is a link to the full dissertation reporting results from this trial — https://scholarworks.uvm.edu/cgi/viewcontent.cgi?article=1922&context=graddis

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Started | 39 | 35
Attended End of Baseline Study Visit | 36 | 32
Completed (Completion defined as attended the final study visit.) | 31 | 27
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Population: The 68 participants who completed baseline were included in the primary analysis. Six participants who were enrolled were not included in the analysis because they withdrew from the study prior to completing baseline or receiving the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (13.4) | 39.3 (13.6) | 38.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 22 | 19 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Six participants (three in each condition) were not included in the analyses because they withdrew from the study before completing baseline or receiving their assigned intervention.
  Participants
    Race/Ethnicity: White, non-Hispanic | 28 | 28 | 56
    Race/Ethnicity: Black, non-Hispanic | 1 | 1 | 2
    Race/Ethnicity: American Indian or Alaska Native, non-Hispanic | 0 | 0 | 0
    Race/Ethnicity: Asian, non-Hispanic | 0 | 0 | 0
    Race/Ethnicity: Pacific Islander, non-Hispanic | 0 | 0 | 0
    Race/Ethnicity: Some other race | 2 | 1 | 3
    Race/Ethnicity: More than one race | 3 | 2 | 5
    Race/Ethnicity: Prefer not to answer | 2 | 0 | 2
    Race/Ethnicity: Hispanic | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Indicated by Self-reported Adherence to Study Cigarettes.
Description: The investigators will use non-adherence to nicotine reduction (i.e., self report of percent non-study cigarettes per day) as an indicator of feasibility.
Time Frame: Assessed weekly during the 4 week reduction period after the baseline week
Population: Feasibility was assessed with percent non-study cigarettes. Greater percent non-study cigarettes per day indicates less feasibility. See the full paper for more detailed outcomes: https://doi.org/10.1111/add.14666
Measure: Mean (Standard Error); unit: Percent non-study cigarettes per day
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Number analyzed (Participants) | 36 | 32
Percent non-study cigarettes per day
  Baseline (Week 0) | 7.1 (0.03) | 7.3 (0.03)
  Week 1 | 10.4 (0.03) | 13.3 (0.04)
  Week 2 | 14.8 (0.05) | 31.2 (0.05)
  Week 3 | 14.1 (0.05) | 52.3 (0.06)
  Week 4 | 21.4 (0.06) | 72.3 (0.06)

2. Primary Outcome: Self Reported Dependence Using the Nicotine Dependence Syndrome Scale (NDSS)
Description: The NDSS is a measure of dependence that does not rely on cigarettes per day as an indicator of dependence.
Time Frame: Assessed weekly during the 4 week reduction period after the baseline week
Population: The NDSS overall score is reported has a t-score (range= -3.9 to 2.3) with lower scores indicating lower nicotine dependence. Please see full paper for further results: https://doi.org/10.1111/add.14666
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Number analyzed (Participants) | 36 | 32
t-score
  Baseline (Week 0) | -0.7 (0.17) | -0.8 (0.18)
  Week 1 | -1.1 (0.15) | -1.0 (0.16)
  Week 2 | -1.2 (0.17) | -1.2 (0.18)
  Week 3 | -1.4 (0.14) | -1.4 (0.15)
  Week 4 | -1.7 (0.15) | -1.3 (0.16)

3. Secondary Outcome: Any Quit Attempt (QA)
Description: The percent of participants in each condition who made one or more self-reported quit attempts to stop smoking for good during the study period, lasting any length of time (including attempts lasting less than 24 hours).
Time Frame: Participants were asked at the end of the reduction period whether they made a quit attempt at any point during the 4 week reduction period.
Measure: Count of Participants; unit: Participants
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Number analyzed (Participants) | 36 | 32
Participants | 6 | 13

4. Secondary Outcome: Number of Participants With Self Reported Seven Day Point Prevalence Abstinence
Description: Self reported seven day point prevalence abstinence.
Time Frame: Assessed at the end of the 4 week reduction period
Measure: Count of Participants; unit: Participants
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Number analyzed (Participants) | 36 | 32
Participants | 0 | 1

5. Secondary Outcome: Self-efficacy to Quit Smoking
Description: Velicer's self-efficacy scale is a self-report measure of self-efficacy to quit smoking (1=least to 5=most).
Time Frame: Week 0 - Week 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
Number analyzed (Participants) | 36 | 32
units on a scale
  Baseline (Week 0) | 2.5 (0.16) | 2.9 (0.17)
  Week 1 | 2.6 (0.17) | 2.7 (0.18)
  Week 2 | 2.7 (0.17) | 2.8 (0.18)
  Week 3 | 3.1 (0.17) | 2.8 (0.19)
  Week 4 | 3.4 (0.18) | 2.6 (0.19)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Switch to VLNC Cigarettes | Reduce CPD
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 30/36 | 25/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to VLNC Cigarettes (N=36) | Reduce CPD (N=32)
Mild chest pain/tightness (General disorders) | 0 (0) | 2 (2)
Mild muscle ache/spasm (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Headache/Dizziness (Investigations) | 3 (4) | 2 (3)
Cough/Mucus (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Heart palpitation (Investigations) | 1 (2) | 1 (1)
Disrupted sleep (Investigations) | 2 (3) | 3 (4)
Mood (Psychiatric disorders) | 3 (4) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Mouth irritation/dryness (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (4)
Other (Investigations) | 4 (4) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03060083/Prot_SAP_001.pdf